CLINICAL TRIAL: NCT04523259
Title: Compatibility Problems and Prescribing Pattern of Injectable Drugs at the Hospital
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200911016R
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: IV Injection
Keywords: Drug incompatibility; injections; infusion, intravenous; medication errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Drug safety is always a national, as well as international, patient safety goal. Administration of injection, especially intravenous infusion, is an extremely complicated and dangerous process, which includes reconstitution, dilution, selection of diluent and volume, verification of concentration of final solution, check for stability, sterility and compatibilities, and the selection of intravenous (IV) set, peripheral or central route, and the rate of infusion. Due to its inherent complexity, errors occur easily during these procedures. Literatures indicated that the incidence of injection administration errors ranged from 13% to 84%, which included errors in dosage, diluents, and volumes; excessive administration rate; and incompatible IV admixture.

In the U.S.A., pharmacists provide comprehensive clinical services. They ensure the appropriateness of every step in the process from prescription and dosage verification, drug reconstitution and dilution, selection of diluents and concentration, to the rate of administration. Even more, they provide the final IV products that are ready to administer to the patients (IV admixture services). Therefore, many common administration errors can be avoided. In Taiwan, nevertheless, pharmacists have limited role in IV services due to our health-care system. There are no studies on the administration pattern of injections. There is still room for improvement in the assurance of injection safety.

To ensure the safety of injection, we not only have to oversee the accuracy of drugs and dosage, but also take the compatibilities among drugs and diluents seriously.

Because diluent is not a mandatory claim data, the National Health Insurance data base cannot provide the related information for drug compatibility epidemiology study. The application for reimbursement of injections is based on total amount used instead of daily usage; it is therefore difficult to find drug incompatibility problems in this data base. Hospital data base analysis, questionnaire survey and chart review are more feasible for such study.

This study will analyze the prescriptions of IV injection in the intensive-care units and pediatric units to determine the prescribing pattern. High risk IV admixtures and Y-site administrations will be explored by questionnaire survey and literature review. Laboratory experiments will be done on some indicator drugs to find the reasons, categories and severities of the compatibilities. A list of incompatible drugs shall be generated for computerized intervention. We hope the results of the study can be used as a reference for guideline, policy and procedure for health care system and government.

ELIGIBILITY:
Inclusion Criteria:

* nurses

Exclusion Criteria:

* not nurses

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: nurse in ICU
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2009-11-09 (Actual); Primary Completion 2010-07-01 (Actual); Study Completion 2013-11-04 (Actual)

PRIMARY OUTCOMES:
Drug incompatibility assessed by questionnaire survey | 6 months
  IV admixture

CONTACTS AND LOCATIONS:
Overall Officials: Taiwan National Taiwan University Hospital, Principal Investigator — National Taiwan University Hospital